CLINICAL TRIAL: NCT05333120
Title: A Clinical Multicenter, Prospective, Observational Cohort Study to Validate a Prediction Mobile APP for Perioperative Hypothermia
Brief Title: Multi-center Validation of a Hypothermia Prediction Mobile Application (APP)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Huang YuGuang, Chief physician, Peking Union Medical College Hospital
Other Study IDs: HypothermiaAPP
Record Dates: First submitted 2022-03-28; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Perioperative Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There have been no fully validated tools for rapid screen of surgical patients at risk of intraoperative hypothermia. The aim of this study is to validate the performance of a previously established prediction model in estimating risk of intraoperative hypothermia using a prospective cohort before further implementation of the model. We hypothesize that the prediction model has helpful discrimination and adequate calibration [1] for clinical use.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational cohort study to validate the property of a previously established mobile application (APP) [2] for estimating risk of intraoperative hypothermia. Patients scheduled for elective surgery under general anesthesia will be enrolled consecutively at 30 hospitals, which are randomly selected across China, between June, 2021 and December 2022. The total planned sample size is 3000 cases. Eligible participants will be identified, informed to sign the consent, and flagged at preoperative interview the day prior to the operation. Anesthetics and perioperative temperature management will be chosen at the discretion of the anesthesiologists without intervention. Intraoperative hypothermia risk score of each participant will be calculated by a mobile application of the predictor model [2] before surgery. A wireless axillary thermometer [3] will be used to continuously measure and record perioperative core temperature as the reference standard. All participants will be followed up until 30 days after the operation.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* undergoing elective operation with general anesthesia or combined with other anesthesia
* operation is expected to last more than 40 minutes

Exclusion Criteria:

* central hyperthermia (e.g., cerebrovascular disease, traumatic brain injury, cerebral operation, epilepsy or acute hydrocephalus)
* impaired thermoregulation (e.g., neuroleptic malignant syndrome, malignant hyperthermia, or known hyperthyroidism/hypothyroidism with current thyroid dysfunction
* infectious fever
* core temperature ≥38.5 ℃ attributable to other causes within 3 days before surgery
* operation with induced hypothermia (e.g. cardiopulmonary bypass)
* unsuited for infrared tympanic thermometry or axillary temperature monitoring
* unwilling to give signed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from 30 hospitals which are randomly selected across China.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
occurrence of perioperative hypothermia | during the perioperative period, an average of 2.5 hours
  core temperature (measured by wireless axillary thermometer) <36.0 ℃ at any time from admission to the preoperative holding area till discharge from post anesthesia care unit (PACU)

SECONDARY OUTCOMES:
amount of blood loss and blood transfusion | during the operation
  amount of blood loss and blood transfusion during the operation
occurrence of shivering and thermal discomfort | during the perioperative period, an average of 2.5 hour
  shivering and thermal discomfort occurring from admission to the preoperative holding area till discharge from post anesthesia care unit (PACU)
duration of hospitalization | during hospitalization, an average of 10 days
  time from hospital admission to hospital discharge
occurrence of myocardial injury non-cardiac surgery (MINS) | during 3 days after the operation
  (1) a non-high-sensitivity troponin T ≥30ng/L, or (2) a high-sensitivity troponin T (hsTnT) ≥65ng/L, or (3) a hsTnT of 20 to <65 ng/L with an absolute change of at least 5 ng/L, or (4) an elevation as any value above the 99th percentile upper reference limit for troponin I [4-6]
occurrence of surgical site infection (SSI) | during 30 days after the operation
  definition of SSI is according to the CDC criterion in 2021 [7]
occurrence of death | during 30 days after the operation
  death occurring in 30 days after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, M.D., Study Chair — Department of Anesthesiology, Peking Union Medical College Hospital
Locations (1):
- Department of Anesthesiology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Alba AC, Agoritsas T, Walsh M, Hanna S, Iorio A, Devereaux PJ, McGinn T, Guyatt G. Discrimination and Calibration of Clinical Prediction Models: Users' Guides to the Medical Literature. JAMA. 2017 Oct 10;318(14):1377-1384. doi: 10.1001/jama.2017.12126. PMID 29049590
- [Background] Yi J, Zhan L, Lei Y, Xu S, Si Y, Li S, Xia Z, Shi Y, Gu X, Yu J, Xu G, Gu E, Yu Y, Chen Y, Jia H, Wang Y, Wang X, Chai X, Jin X, Chen J, Xu M, Xiong J, Wang G, Lu K, Yu W, Lei W, Qin Z, Xiang J, Li L, Yao M, Huang Y. Establishment and Validation of a Prediction Equation to Estimate Risk of Intraoperative Hypothermia in Patients Receiving General Anesthesia. Sci Rep. 2017 Oct 24;7(1):13927. doi: 10.1038/s41598-017-12997-x. PMID 29066717
- [Background] Pei L, Huang Y, Mao G, Sessler DI. Axillary Temperature, as Recorded by the iThermonitor WT701, Well Represents Core Temperature in Adults Having Noncardiac Surgery. Anesth Analg. 2018 Mar;126(3):833-838. doi: 10.1213/ANE.0000000000002706. PMID 29293176
- [Background] Botto F, Alonso-Coello P, Chan MT, Villar JC, Xavier D, Srinathan S, Guyatt G, Cruz P, Graham M, Wang CY, Berwanger O, Pearse RM, Biccard BM, Abraham V, Malaga G, Hillis GS, Rodseth RN, Cook D, Polanczyk CA, Szczeklik W, Sessler DI, Sheth T, Ackland GL, Leuwer M, Garg AX, Lemanach Y, Pettit S, Heels-Ansdell D, Luratibuse G, Walsh M, Sapsford R, Schunemann HJ, Kurz A, Thomas S, Mrkobrada M, Thabane L, Gerstein H, Paniagua P, Nagele P, Raina P, Yusuf S, Devereaux PJ, Devereaux PJ, Sessler DI, Walsh M, Guyatt G, McQueen MJ, Bhandari M, Cook D, Bosch J, Buckley N, Yusuf S, Chow CK, Hillis GS, Halliwell R, Li S, Lee VW, Mooney J, Polanczyk CA, Furtado MV, Berwanger O, Suzumura E, Santucci E, Leite K, Santo JA, Jardim CA, Cavalcanti AB, Guimaraes HP, Jacka MJ, Graham M, McAlister F, McMurtry S, Townsend D, Pannu N, Bagshaw S, Bessissow A, Bhandari M, Duceppe E, Eikelboom J, Ganame J, Hankinson J, Hill S, Jolly S, Lamy A, Ling E, Magloire P, Pare G, Reddy D, Szalay D, Tittley J, Weitz J, Whitlock R, Darvish-Kazim S, Debeer J, Kavsak P, Kearon C, Mizera R, O'Donnell M, McQueen M, Pinthus J, Ribas S, Simunovic M, Tandon V, Vanhelder T, Winemaker M, Gerstein H, McDonald S, O'Bryne P, Patel A, Paul J, Punthakee Z, Raymer K, Salehian O, Spencer F, Walter S, Worster A, Adili A, Clase C, Cook D, Crowther M, Douketis J, Gangji A, Jackson P, Lim W, Lovrics P, Mazzadi S, Orovan W, Rudkowski J, Soth M, Tiboni M, Acedillo R, Garg A, Hildebrand A, Lam N, Macneil D, Mrkobrada M, Roshanov PS, Srinathan SK, Ramsey C, John PS, Thorlacius L, Siddiqui FS, Grocott HP, McKay A, Lee TW, Amadeo R, Funk D, McDonald H, Zacharias J, Villar JC, Cortes OL, Chaparro MS, Vasquez S, Castaneda A, Ferreira S, Coriat P, Monneret D, Goarin JP, Esteve CI, Royer C, Daas G, Chan MT, Choi GY, Gin T, Lit LC, Xavier D, Sigamani A, Faruqui A, Dhanpal R, Almeida S, Cherian J, Furruqh S, Abraham V, Afzal L, George P, Mala S, Schunemann H, Muti P, Vizza E, Wang CY, Ong GS, Mansor M, Tan AS, Shariffuddin II, Vasanthan V, Hashim NH, Undok AW, Ki U, Lai HY, Ahmad WA, Razack AH, Malaga G, Valderrama-Victoria V, Loza-Herrera JD, De Los Angeles Lazo M, Rotta-Rotta A, Szczeklik W, Sokolowska B, Musial J, Gorka J, Iwaszczuk P, Kozka M, Chwala M, Raczek M, Mrowiecki T, Kaczmarek B, Biccard B, Cassimjee H, Gopalan D, Kisten T, Mugabi A, Naidoo P, Naidoo R, Rodseth R, Skinner D, Torborg A, Paniagua P, Urrutia G, Maestre ML, Santalo M, Gonzalez R, Font A, Martinez C, Pelaez X, De Antonio M, Villamor JM, Garcia JA, Ferre MJ, Popova E, Alonso-Coello P, Garutti I, Cruz P, Fernandez C, Palencia M, Diaz S, Del Castillo T, Varela A, de Miguel A, Munoz M, Pineiro P, Cusati G, Del Barrio M, Membrillo MJ, Orozco D, Reyes F, Sapsford RJ, Barth J, Scott J, Hall A, Howell S, Lobley M, Woods J, Howard S, Fletcher J, Dewhirst N, Williams C, Rushton A, Welters I, Leuwer M, Pearse R, Ackland G, Khan A, Niebrzegowska E, Benton S, Wragg A, Archbold A, Smith A, McAlees E, Ramballi C, Macdonald N, Januszewska M, Stephens R, Reyes A, Paredes LG, Sultan P, Cain D, Whittle J, Del Arroyo AG, Sessler DI, Kurz A, Sun Z, Finnegan PS, Egan C, Honar H, Shahinyan A, Panjasawatwong K, Fu AY, Wang S, Reineks E, Nagele P, Blood J, Kalin M, Gibson D, Wildes T; Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Writing Group, on behalf of The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Investigators; Appendix 1. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Study Investigators Writing Group; Appendix 2. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN Operations Committee; Vascular events In noncardiac Surgery patIents cOhort evaluatioN VISION Study Investigators. Myocardial injury after noncardiac surgery: a large, international, prospective cohort study establishing diagnostic criteria, characteristics, predictors, and 30-day outcomes. Anesthesiology. 2014 Mar;120(3):564-78. doi: 10.1097/ALN.0000000000000113. PMID 24534856
- [Background] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280
- [Background] Devereaux PJ, Szczeklik W. Myocardial injury after non-cardiac surgery: diagnosis and management. Eur Heart J. 2020 May 1;41(32):3083-3091. doi: 10.1093/eurheartj/ehz301. PMID 31095334
- [Background] National Healthcare Safety Network, Centers for Disease Control and Prevention. Surgical site infection (SSI) event. http://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf. Published January 2021. Accessed May 21, 2021.